CLINICAL TRIAL: NCT01774149
Title: Data Driven Feedback as a Method to Improve Glycaemic Control in Type 1 Diabetes
Brief Title: Model Driven Diabetes Care
Acronym: MDDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011/1939 (REK)
Record Dates: First submitted 2013-01-11; First posted 2013-01-23 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Diastat (Active Comparator): Mobile phone application Few Touch Application (FTA) in the regular version, with Diastat turned on in week 12 post-enrollment.
  Interventions: Device: Few Touch Application; Device: Diastat
- Diastat (Experimental): Few Touch Application with Diastat module turned on in week 4 post-enrollment.
  Interventions: Device: Few Touch Application; Device: Diastat

INTERVENTIONS:
Device: Few Touch Application — Users get access to the regular version of the Few Touch Application for Type 1 Diabetes.
  Other Names: Diabetesdagboka
Device: Diastat — Users get the Few Touch Application with Diastat module activated.

SUMMARY:
Patients with Diabetes Mellitus Type 1 using electronic self-help tools typically registers a large amount of data on their disease. The study intends to see if giving advanced feedback on these data can improve their blood glucose management.

DETAILED DESCRIPTION:
All patients will be given access to a mobile phone with the diabetes diary known as the Few Touch Application (FTA) installed. They may use either their own compatible Android handsets, or provided handsets. The study uses a delayed start design. Participants are randomized into two groups, who get access to the module "Diastat" after 4 and 12 weeks post-enrollment respectively. Each group uses the FTA with Diastat for 8 weeks post-intervention (i.e. access to Diastat).

Diastat is a module within FTA that provides data-driven feedback to the patients using their own data. This module is based on the data recorded in a previous trial [1]. Three submodules are part of Diastat; Periodicity detection and visualization, multiscale trend detection based on the c-SiZer algorithm [2], and situation matching for insulin dosage [3].

1. Skrøvseth SO et al, Diabetes Technol Ther (2012)
2. Skrøvseth SO et al, PLoS ONE (2012)
3. Skrøvseth SO et al, Accepted for Advanced Technologies and Treatments for Diabetes, Paris, France, 2013.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis with Diabetes Mellitus type 1 for at least one year.
* Age over 18 years
* Has basic familiarity with mobile phones, and uses mobile phone on a daily basis.

Exclusion Criteria:

* Severe complications due to their diabetes.
* Unable to understand or conform to the guidelines when presented with the phone's software.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stein Olav Skrøvseth, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hopital of North Norway, Tromsø, Norway

REFERENCES:
- [Background] Skrovseth SO, Arsand E, Godtliebsen F, Hartvigsen G. Mobile phone-based pattern recognition and data analysis for patients with type 1 diabetes. Diabetes Technol Ther. 2012 Dec;14(12):1098-104. doi: 10.1089/dia.2012.0160. Epub 2012 Oct 4. PMID 23035775
- [Background] Skrovseth SO, Arsand E, Godtliebsen F, Joakimsen RM. Model driven mobile care for patients with type 1 diabetes. Stud Health Technol Inform. 2012;180:1045-9. PMID 22874353
- [Background] Arsand E, Froisland DH, Skrovseth SO, Chomutare T, Tatara N, Hartvigsen G, Tufano JT. Mobile health applications to assist patients with diabetes: lessons learned and design implications. J Diabetes Sci Technol. 2012 Sep 1;6(5):1197-206. doi: 10.1177/193229681200600525. PMID 23063047
- [Background] Skrovseth SO, Bellika JG, Godtliebsen F. Causality in scale space as an approach to change detection. PLoS One. 2012;7(12):e52253. doi: 10.1371/journal.pone.0052253. Epub 2012 Dec 27. PMID 23300626
- [Background] Skrovseth SO, Arsand E, Godtliebsen F, Joakimsen RM. Model-driven diabetes care: study protocol for a randomized controlled trial. Trials. 2013 May 14;14:139. doi: 10.1186/1745-6215-14-139. PMID 23672413
- [Derived] Skrovseth SO, Arsand E, Godtliebsen F, Joakimsen RM. Data-Driven Personalized Feedback to Patients with Type 1 Diabetes: A Randomized Trial. Diabetes Technol Ther. 2015 Jul;17(7):482-9. doi: 10.1089/dia.2014.0276. Epub 2015 Mar 9. PMID 25751133

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Delayed Diastat | Diastat
Started | 15 | 15
Completed | 14 | 12
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Diastat | Diastat | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (7.3) | 41.1 (13.5) | 39.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  Norway | 15 | 15 | 30
HbA1c [Mean (Standard Deviation); unit: %] | 8.06 (1.32) | 8.33 (0.87) | 8.20 (1.11)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Frequency of Hyper- and Hypo-glycemic Events From Baseline to Week 8-12.
Description: The number of self-measured blood glucose values < 4 mmol/L (72 mg/dL) or > 15 mmol/L (270 mg/dL) will be recorded during baseline (first 4 weeks post-enrollment/start of study) and during weeks 8-12 post-enrollment for all participants.
Time Frame: Up to 12 weeks post-enrollment
Population: 14 participants in each group were active users and had sufficient data to be analyzed for the outcome.
Measure: Mean (95% Confidence Interval); unit: Events
Arm/Group | Delayed Diastat | Diastat
Number analyzed (Participants) | 14 | 14
Events | -18 [-25 to -13] | -7.5 [-15.5 to -.5]

2. Secondary Outcome: Change in HbA1c
Description: HbA1c will be measured at the start of the study (week 1 post-enrollment) and during the last week of intervention (week 12 for the intervention group and week 20 for the active comparator group).
Time Frame: up to 20 weeks post-enrollment
Population: 11 participants in each group met for measurement of HbA1c. Reasons for not meeting was not recorded.
Measure: Mean (95% Confidence Interval); unit: Percentage points
Arm/Group | Delayed Diastat | Diastat
Number analyzed (Participants) | 11 | 11
Percentage points | -0.57 [-1.1 to -.05] | -0.63 [-1.02 to -0.24]

3. Other Pre Specified Outcome: Usability
Description: System Usability Scale (SUS) will be applied to assess usability of the approach and recorded during the last week of intervention (week 12 for the intervention group and week 20 for the active comparator group).
Time Frame: up to 20 weeks post-enrollment
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Empowerment
Description: Diabetes Empowerment Scale-Short Form (DES-SF) will be used to assess empowerment at the start of the study (week 1 post-enrollment) and during week 12 of intervention.
Time Frame: Up to 12 weeks post-enrollment.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Delayed Diastat | Diastat
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No